CLINICAL TRIAL: NCT07309419
Title: A Prospective, Randomized, Open-Label, Multicenter Phase III Trial Evaluating the Efficacy and Safety of Transarterial Chemoembolization Combined With an Oral Triple-Agent Cocktail Regimen Versus Transarterial Chemoembolization Combined With First-Line Targeted Therapy Plus Immunotherapy in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: A Phase III Randomized Study of TACE Plus an Oral Triple-Agent Cocktail Versus TACE Plus First-Line Targeted Immunotherapy in Unresectable Hepatocellular Carcinoma
Acronym: Cocktail-001
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jinglin Xia, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2025-745R
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib; camrelizumab; Thalidomide; Pharmaceutical Preparations; Capecitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: apatinib + camrelizumab + TACE (Active Comparator): Participants will receive apatinib plus camrelizumab on Day 1 of a 21-Day cycle, after every on-demand transarterial chemoembolization procedure.
  Interventions: Drug: Apatinib; Drug: Camrelizumab; Device: TACE
- Arm B: Thalidomide + Capecitabine + Compound cantharides capsule + TACE (Experimental): Participants assigned to this arm will receive an oral triple-agent regimen consisting of thalidomide, capecitabine, and compound cantharides capsules. The oral regimen will be initiated immediately after the initial transarterial chemoembolization (TACE) procedure and administered continuously thereafter.
  Interventions: Device: TACE; Drug: Thalidomide (drug); Drug: Capecitabine; Drug: Compound cantharides capsule

INTERVENTIONS:
Drug: Apatinib — Apatinib: 250m, po, QD
  Arms: Arm A: apatinib + camrelizumab + TACE
Drug: Camrelizumab — Camrelizumab: 200mg, iv, Q3W
  Arms: Arm A: apatinib + camrelizumab + TACE
Device: TACE — TACE if necessary
Drug: Thalidomide (drug) — Thalidomide：50-75mg, PO, qn;
  Arms: Arm B: Thalidomide + Capecitabine + Compound cantharides capsule + TACE
Drug: Capecitabine — Capecitabine: 500mg, PO, bid
  Arms: Arm B: Thalidomide + Capecitabine + Compound cantharides capsule + TACE
Drug: Compound cantharides capsule — Compound cantharides capsule: 750mg, PO, tid
  Arms: Arm B: Thalidomide + Capecitabine + Compound cantharides capsule + TACE

SUMMARY:
This is a prospective, multicenter, randomized, open-label phase 3 study evaluating the efficacy and safety of transarterial chemoembolization (TACE) combined with a triple oral cocktail regimen versus TACE combined with targeted therapy plus immunotherapy as first-line treatment for unresectable hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of enrollment.
* Diagnosis of hepatocellular carcinoma (HCC) established according to the Chinese National Liver Cancer (CNLC) guidelines, based on imaging findings and/or histopathological confirmation.
* Not eligible for curative treatment, including surgical resection, local ablation, or liver transplantation.
* No prior treatment for HCC, including any locoregional or systemic anticancer therapies.
* Child-Pugh liver function class A or B 7.

Exclusion Criteria:

* Participants who had another previous or current malignant tumor, except for early-stage cancer with low risk of recurrence or a malignant tumor curatively treated >5 years prior to enrolment with no recurrence
* Participants who have severe allergy to iodine, and unable to receive TACE
* Participants who have undergone a liver transplant or allogeneic bone marrow transplantation, or those who are in the waiting list for liver or bone marrow transplantation
* Participants who had congenital or acquired immune deficiency, such as HIV infection
* Participants who had a history of gastrointestinal bleeding within 6 months prior to randomization or a definite tendency of gastrointestinal bleeding
* Participants who had undergone arterial thromboembolism within 6 months prior to randomization or a definite tendency of gastrointestinal bleeding, such as cerebrovascular accident, ≥ CTCAE grade 3 deep vein thrombosis and pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to ~4 years
  Overall survival is defined as the time from randomization to death from any cause. OS will be assessed in the intention-to-treat (ITT) population, which includes all randomized participants.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to ~2 years
  Progression-free survival is defined as the time from randomization to the first documented disease progression or death from any cause, whichever occurs first. Tumor progression will be assessed according to the RECICL criteria and the mRECIST criteria by investigators and a blinded independent radiology committee (BIRC) in the ITT population.
Time to Progression (TTP) | Up to ~2 years
  Time to progression is defined as the time from randomization to disease progression that is no longer amenable to transarterial chemoembolization (TACE failure or refractoriness), as assessed according to RECICL and mRECIST criteria in the ITT population.
Objective Response Rate (ORR) | Up to ~2 years
  Objective response rate is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) after treatment initiation. Tumor response will be assessed according to RECICL and mRECIST criteria by investigators and the BIRC in the ITT population.
Duration of Response (DOR) | Up to ~2 years
  Duration of response is defined as the time from the first documented CR or PR to disease progression or death from any cause, whichever occurs first. DOR will be assessed according to RECICL and mRECIST criteria in the ITT population.
Health-Related Quality of Life (HRQoL) | Up to ~2 years
  Health-related quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).

IPD SHARING:
Plan to Share IPD: No